CLINICAL TRIAL: NCT01241045
Title: EFFECT OF VAGINAL Ph AND ACIDIFICATION OF VAGINAL MISOPROSTOL ON ITS EFFICACY FOR INDUCTION OF MID-TRIMESTERIC ABORTION
Brief Title: Study of Effect of Vaginal ph and Acidification of Vaginal Misoprostol on Its Efficacy for Induction of Midtrimester Abortion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Ain Shams University, Ain Shams University
Other Study IDs: AubshamsU
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: To Evaluate the Impact of the Vaginal Ph and Acidification of Vaginal Misoprostol on Its Efficacy in Facilitating Induction of Mid-trimester Abortion.

STUDY DESIGN:
Observational Model: Ecologic or Community
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- misoprostol: 2 groups:-
  * Group 1:-those with Ph<5. (n=50).
  * Group 2:-those with Ph > or=5. (n=50). -Each group is subdivided into another two groups:-
    * Group 1A (n=25). - Group 1B (n=25).
    * Group 2A (n=25). - Group 2B (n=25).
    * All the women in group 1A and group 2A will receive intravaginal misoprostol tablets moistened with 3 ml of 5% acetic acid, and all the women in group 1B and group 2B will receive intravaginal misoprostol tablets moistened with water, 400 micrograms every 4 hours for a maximum of 5 doses within 24 hours. If the patient will not have adequate uterine contractions, the same regimen will be repeated over the following 24 hours

SUMMARY:
To evaluate the impact of the vaginal Ph and acidification of vaginal misoprostol on its efficacy in facilitating induction of midtrimester abortion.

DETAILED DESCRIPTION:
100 Pregnant women, in mid-trimester, with a medical indication for termination of pregnancy will be approached to participate in this study Methods:-

1. A formal consent from the women under study with full notification and explanation of the methods, importance of the study and possible unwanted effects.
2. During the pre-selection visit, exclusion and inclusion criteria will be applied. Baseline investigations; Blood sugar, Serum Glutamate Oxaloacetate Transaminase (SGOT), Serum Glutamate Pyruvate Transaminase (SGPT), S. Creatinine, and Complete Blood Count (C.B.C.) and Coagulation profile (PTT, serum fibrinogen level) will be done.
3. Following admission, all patients will undergo complete clinical examination and detailed medical history will be obtained. Each patient will have a Case Record Form (CRF) in which the following data will be recorded.

   * Patient initials.
   * Patient number (according to the randomization schedule).
   * Age, height, weight,
   * Known allergies.
   * Past medical and surgical history (no longer present).
   * Medications taken within the last 4 weeks and discontinued.
   * Concomitant illnesses.
   * Concomitant medications which will not be discontinued.
   * Clinical examination: including full gynaecologic assessment including vaginal and speculum examination with recording of vaginal and cervical condition.
4. The vaginal Ph will be measured using Universal indicator paper pH (1-14) before digital vaginal examination. Through speculum examination, the indicator will be held with an artery forceps against the vaginal wall-high up in the vagina-until it becomes wet.

   Color change of the strip will be immediately compared with the colorimetric scale and the measurement will be recorded.

   Patients will be divided into 2 groups:-
   * Group 1:-those with Ph<5. (n=50).
   * Group 2:-those with Ph > or=5. (n=50).
5. Each group is subdivided into another two groups:-

   * Group 1A (n=25). - Group 1B (n=25).
   * Group 2A (n=25). - Group 2B (n=25).
6. All the women in group 1A and group 2A will receive intravaginal misoprostol tablets moistened with 3 ml of 5% acetic acid, and all the women in group 1B and group 2B will receive intravaginal misoprostol tablets moistened with water, 400 micrograms every 4 hours for a maximum of 5 doses within 24 hours. If the patient will not have adequate uterine contractions, the same regimen will be repeated over the following 24 hours, and if no response will be achieved, this will be considered a failure of therapy, and another method will be used like large doses of oxytocin or cervical dilatation by foley's catheter no.16.
7. assessment will be though the occurrence of uterine contraction and progress of abortion with induction -termination interval as a primary outcome.
8. The investigator will supervise application of the medication dose by dose. Subjects withdrawn from the study before the onset of spontaneous labor

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:-

  1. Age 18-45 years.
  2. A valid indication for termination of pregnancy.
  3. Singleton pregnancy.
  4. Gestational age ranging between 14 and 26 weeks of pregnancy.
  5. Uterus and cervix are apparently normal on clinical examination.
  6. Cervix is not dilated with absence of effacement.
  7. Absence of uterine activity.
  8. Written and signed informed consent by the patient to participate in the study.

Exclusion Criteria:

* Exclusion Criteria:-

  1. A contraindication to medical termination of pregnancy e.g. placenta praevia.
  2. Evidences suggesting onset of spontaneous abortion (uterine contractions with or without cervical changes).
  3. Previous trial to induce abortion or the use of pre-induction agent during the current pregnancy.
  4. Any contraindication to receiving prostaglandins, including known hypersensitivity to misoprostol or other prostaglandins (PGs), history of asthma, glaucoma, cardiac or cardiovascular disease.
  5. Parity six or more.
  6. Multifetal pregnancy.
  7. Severe Polyhydramnios.
  8. Presence of vaginal bleeding.
  9. Presence of ruptured membranes and/or suspicion of septic abortion as evidenced by maternal temperature of 38°C or more, uterine tenderness or foul-smelling vaginal discharge.
  10. Previous Caesarean section or other uterine surgery or perforation.
  11. Cervical cerclage during current pregnancy, or history of it during a previous pregnancy.
  12. Previous cervical surgery as cauterization of cervical erosion or cervical dilatation operation with resultant apparent cervical tears or lacerations.
  13. Metabolic acidosis as a result of a medical disorder.
  14. Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol which include all vaginal forms of medications.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
induction-termination interval | 11 hours
  time elapsed from admenstiration of drug to occurrence of abortion

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams, Cairo, California, United States